CLINICAL TRIAL: NCT03874793
Title: Neural Mechanisms of Mindfulness-based Cognitive Therapy (MBCT) for Posttraumatic Stress Disorder (PTSD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); University of Michigan (Other)
Responsible Party: Principal Investigator, Anthony P King, Associate Professor of Psychiatry and Behaviroal Health, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00152509; 1R61AT009867-01 (NIH)
Record Dates: First submitted 2019-03-12; First posted 2019-03-14 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Mindfulness-Based Cognitive Therapy; Muscle Relaxation; fMRI; Group Psychotherapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Intervention Model Description: treatment groups will consist of a minimum of 4 participants (preferably 5-8). The statistician will randomize the groups once a sufficient number of participants have enrolled to ensure desired group size.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Statistician will not know the group assignment until blind is broken. Statistician randomizes the groups. Principal investigator will not know group assignment until blind is broken.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Cognitive Therapy (Experimental): Participants will have 8 weeks of group therapy and will be asked to do MBCT exercises for approximately 20-30 minutes on 5 or more days/week.
  Interventions: Behavioral: Mindfulness-Based Cognitive Therapy
- Muscle Relaxation Therapy (MRG) (Active Comparator): Participants will have 8 weeks of group therapy participants and will be asked to do MRG exercises for approximately 20-30 minutes on 5 or more days/week.
  Interventions: Behavioral: Muscle Relaxation Therapy

INTERVENTIONS:
Behavioral: Mindfulness-Based Cognitive Therapy — Participants will attend 8 weekly group therapy sessions. Prior to and after therapy participants will have assessments related to their PTSD, fill out surveys, and have an fMRI.
  Arms: Mindfulness-Based Cognitive Therapy
Behavioral: Muscle Relaxation Therapy — Participants will attend 8 weekly group therapy sessions. Prior to and after therapy participants will have assessments related to their PTSD, fill out surveys, and have an fMRI.
  Arms: Muscle Relaxation Therapy (MRG)

SUMMARY:
This study will examine the effects of psychotherapy as treatment for PTSD, and specifically how brain activity and brain connectivity is affected by Mindfulness Based Cognitive Therapy (MBCT) and an active mind-body comparison comparison therapy.

DETAILED DESCRIPTION:
This research will see how brain activity and brain connectivity is affected by Mindfulness Based Cognitive Therapy (MBCT) and an active comparison therapy called Muscle Relaxation Therapy (MRT). Participants that qualify to be in this study will be randomly assigned to receive 8 weeks of group therapy in either MBCT or MRT treatments. Prior to receiving therapy participants will: complete baseline assessments related to their PTSD; fill out surveys; have an functional magnetic resonance imaging (fMRI); and provide saliva samples. These assessments will be repeated after the therapy is over. Overall study participation should last approximately 10-12 weeks.

Due to COVID precautions, treatments shifted from in-person to remotely-delivered ("Zoom" video-conferencing) modality.

ELIGIBILITY:
Inclusion Criteria:

* Meets current Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-5) criteria for PTSD (with or without Major Depressive Disorder) or subsyndromal PTSD (has qualifying trauma, has intrusive and avoidant symptoms, and at least one negativity and one arousal symptom, and significant impairment); type of trauma shall be interpersonal violence, combat, and/or sexual assault, etc.

Exclusion Criteria:

* Dissociative PTSD
* Delayed-onset PTSD
* Magnetic Resonance Imaging (MRI) contraindications (e.g. metal in body, inability to be in the scanner - claustrophobia, severe back pain, etc.)
* Serious medical or neurologic conditions (e.g. stroke, seizures)
* Suicide risk
* Psychosis
* Life history of schizophrenia
* Life history of bipolar disorder
* Current substance dependence
* Other factors that preclude safe and meaningful participation in the study, at discretion of the PI and study team

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Group differences in the change in resting-state functional connectivity between posterior cingulate cortex (PCC) and dorsolateral prefrontal cortex (dlPFC) | pre-therapy and post therapy (approximately 8 weeks)
  Network functional connectivity will be measured through fMRI blood oxygen level dependent [BOLD] signal. Time-course of BOLD signal while participants are "resting" / not performing a task will be used identify brain regions whose activity time-course is correlated with a brain region of interest (ROI), called a "seed" ROI. We will use activity in the PCC as a seed ROI and search for regions of time-course correlation within the dlPFC, searching for dlPFC clusters within an anatomical mask of middle frontal cortex. Betas for identified dlPFC clusters will be extracted.

SECONDARY OUTCOMES:
Group differences in the change in resting-state functional connectivity between posterior cingulate cortex (PCC) and insular cortex (Ins) | pre-therapy and post therapy (approximately 8 weeks)
  Network functional connectivity will be measured through fMRI BOLD signal. Time-course of BOLD signal while participants are "resting" / not performing a task will be used identify brain regions whose activity time-course is correlated with a PCC seed ROI and search for regions of time-course correlation within the insula cortex, searching for clusters within an anatomical mask of insular cortex. Betas for identified insula clusters will be extracted.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony King, Ph.D., Principal Investigator — Ohio State University; David Fresco, Ph.D, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes
We plan to make available data from fMRI scans from human subjects initially to collaborators for independent replication / data pooling. We also plan to make the de-identified brain scans available to the broad scientific community, however, additional redaction steps may need to be made to brain scans to ensure subject confidentiality / inability to identify individuals from brain scans. Completely de-identified research data (redacted according to NIH practice to prevent disclosure of personal identifiers) which documents the research findings will be made available after the main findings from the finalized research dataset have been accepted for publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 36 months of completion of the project.
Access Criteria: Access to data generated by the project will be available for educational, research and non-profit purposes to researchers who provide a methodologically sound proposal. Data generated under this project will be administered in accordance with NIH Sharing policies, including NIH Policy on Dissemination of NIH-Funded Clinical Trial Information (8/2016), and the NIH Grants Policy Statement (Availability of Research Results) (11/2015). Depending on such NIH policies, Data generated by this project may be available for educational, research or non-commercial purposes under the terms of a data use agreement. Data will be stored in an established data repository (e.g. Inter-university Consortium for Political and Social Research (ICPSR): icpsr.umich.edu) with appropriate provisions for curation and longterm preservation.